CLINICAL TRIAL: NCT07401264
Title: Multicenter Prospectively Collected Registry of Images and Videos of Colonic Lesions to Develop Artificial Intelligence to Predict Submucosal Invasion
Brief Title: Prospective Image Collection of Colorectal Polyps.
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof. Dr. Raf Bisschops, Prof. Dr., Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S65253
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-09

CONDITIONS: Colonic Lesions
Keywords: image registry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It concerns a study in which we wish to collect images and corresponding histological information (microscopic characteristics) in a prospective manner in various European and non-European centers (multicentric). This means that the collection of images is new and happens in the context of a procedure that has not yet been carried out. The relevant procedure will involve a standard colonoscopy during which we wish to collect digital images and videos of large colorectal polyps (colorectal lesions). These images will later be used for the development of a new computer software (artificial intelligence) that is able to predict the histology (microscopic characteristics) and extent of invasion in the intestinal wall (submucosal invasion) all by itself. The latter is one of the goals in the European project ECOPOP in which the sponsor is involved.

ELIGIBILITY:
Inclusion Criteria:

* Referral for standard or therapeutic colonoscopy
* Digital video material of standard colonoscopy containing at least one colorectal polyp (≥ 10mm) and/or with suspicion of malignancy/submucosal invasion
* Digital images of colorectal polyps ≥ 10mm made during standard colonoscopy and/or with suspicion of malignancy/submucosal invasion Page 11 of 21
* Videos and/or images can be made in white light or any virtual of dye-based enhancement technique
* Colonoscopies performed after IRB approval for this particular study.
* Material collected in adult patients of all sex or race, including pregnant women.

Exclusion Criteria:

* Any contraindication to undergo a standard colonoscopy
* Any uncontrolled coagulopathy or bleeding disorder
* Colonoscopy videos not containing any or colorectal polyps < 10mm
* Colonoscopy videos or images of low quality due to unstable imaging, stool remnants, bowel or patient movements or blurry vision
* Colonoscopy videos with visualization of the polyp less than 5 seconds due to unstable positioning, passing stool remnants, bowel or patient movements or blurry visions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients who need a standard or therapeutic colonoscopy
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-04-07 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
registry of images of colonic lesions | 5 year

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium